CLINICAL TRIAL: NCT02035774
Title: A Novel Selective Block of the Suprascapular Nerve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Lars Marius Ytrebo, Professor, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSNB
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Ligament Injury; Fracture
Keywords: Brachial plexus block; Suprascapular nerve block
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LSIB +SSNB (Active Comparator): Patients will receive LSIB (31 ml ropivacaine 7.5 mg/ml)+ SSNB (4 ml Ropivacaine 5 mg/ml)
  Interventions: Procedure: LSIB + SSNB
- LSIB + placebo (Placebo Comparator): Patients will receive LSIB (31 ml ropivacaine 7.5 mg/ml) + SSNB (4 ml saline)
  Interventions: Procedure: LSIB + SSNB

INTERVENTIONS:
Procedure: LSIB + SSNB — Patients will receive LSIB (31 ml ropivacaine 7.5 mg/ml)+ SSNB (4 ml Ropivacaine 5 mg/ml) or LSIB (31 ml ropivacaine 7.5 mg/ml)+ SSNB (4 ml placebo, saline)

SUMMARY:
Patients who receive the lateral and sagittal infraclavicular block (LSIB) tend to supinate their hand and forearm which may hamper optimal positioning for surgery of the dorsal side of the hand. The investigators think that this supination is caused by lateral rotation in the shoulder. The main lateral rotator of the shoulder is the infraspinatus muscle, which is innervated by the suprascapular nerve (SSN).The investigators hypothesized that optimal positioning of the hand for surgery on the dorsal side of the hand may be achieved by performing a SSN block (SSNB) in addition to the LSIB.

DETAILED DESCRIPTION:
According to the hypothesis the investigators will perform a double blind , placebo controlled study to answer the research question above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists physical status (ASA) I- III
* age between 18 and 70 years
* body mass index between 20 and 36 kg/m2 scheduled for elective hand surgery.

Exclusion Criteria:

We will measure the angle between wrist and horizontal plane while the patient is supine and the extended arm 75° abducted.

* Patient who are not able to pronate the hand ≤15° before block performance, will be excluded from the study.
* Patients will also be excluded if they are pregnant, have contraindications to regional anesthesia, coagulation disorder, allergy to local anesthetics (LA), atrioventricular block, peripheral neuropathy or drug-treated diabetes.
* Patients using other anticoagulation drugs than acetylsalicylic acids or dipyridamol will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Wrist angle | 30 minutes
  The investigators will assess the wrist angle 30 minutes after the two blocks (LSIB + SSNB)

SECONDARY OUTCOMES:
Satisfaction score | 3 hours
  The investigators will ask the surgeons about his/her satisfaction with the hand position during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lars M Ytrebø, Professor, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

REFERENCES:
- [Background] Hackworth RJ. A new and simplified approach to target the suprascapular nerve with ultrasound. J Clin Anesth. 2013 Jun;25(4):347-8. doi: 10.1016/j.jclinane.2013.01.006. Epub 2013 May 1. No abstract available. PMID 23643887
- [Background] Siegenthaler A, Moriggl B, Mlekusch S, Schliessbach J, Haug M, Curatolo M, Eichenberger U. Ultrasound-guided suprascapular nerve block, description of a novel supraclavicular approach. Reg Anesth Pain Med. 2012 May-Jun;37(3):325-8. doi: 10.1097/AAP.0b013e3182409168. PMID 22222688